CLINICAL TRIAL: NCT03432962
Title: Brand Level Nutrient Information Compared to Generic Food Codes: Impact on Results From Dietary Recalls
Brief Title: Brand Level Nutrient Information Compared to Generic Food Codes
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: British Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Janet Cade, Professor of Nutritional Epidemiology, University of Leeds
Other Study IDs: NEG1
Record Dates: First submitted 2018-01-18; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Diet Records; Diet Surveys

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Food code group: The participants freely selected foods from the online dietary assessment tool to record what they had eaten over the last 24h. They then provided information on brand details. The recalls were recoded to take into account all branded items and then recoded again to take represent all generic (ie. no brands) foods.
  Interventions: Other: no intervention - recoding of food recall only

INTERVENTIONS:
Other: no intervention - recoding of food recall only — recoding of food recall

SUMMARY:
Measuring diet is difficult. This is the first time that brand level foods and nutrient values have been compared with generic food codes to explore the difference this might make to estimated nutrient intakes.

DETAILED DESCRIPTION:
Background Traditional dietary assessment methods lack precision. myfood24 is an online 24-hour dietary assessment tool, aiming to reduce the burden of dietary assessment; providing data entry by participants using automated coding of food items. myfood24 includes a large branded food database.

Objective To assess the effect of using brand level nutrient information compared to generic food codes on estimated nutrient intakes.

Design A 24 hour recall was collected using myfood24, which contains a food and nutrient database of over 40,000 items with both branded and generic foods. Participants freely selected their foods generating the 'free choice recall'. After the online recall was completed, they provided further details of brands consumed. The free choice recalls were recoded forming an 'all branded' and an 'all generic' recall. Estimated nutrient intakes from the three different methods of food coding were compared to assess the impact of brand-level information.

ELIGIBILITY:
Inclusion Criteria:

* students University of Leeds
* convenience sample of general public
* adults

Exclusion Criteria:

* none defined

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In order to reach a broad range of individuals, adult participants from both the University of Leeds and from a convenience sample of members of the public, were invited to participate in the study via email.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Nutrient intakes by food coding | 24hour recall
  comparison of nutrient intakes as a result of the recoding process with brand level data

CONTACTS AND LOCATIONS:
Locations (1):
- Nutritional Epidemiology Group, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No